CLINICAL TRIAL: NCT02225522
Title: Prospective Randomized Trial of the Clinical Utility of Rapid Next Generation Sequencing in Acutely Ill Neonates
Brief Title: Genomic Sequencing in Acutely Ill Neonates
Acronym: NSIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HD13-010
Record Dates: First submitted 2014-08-13; First posted 2014-08-26 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2016-09

CONDITIONS: Diseases/Diagnoses; Genetic Disease
Keywords: Intensive Care Units, Neonatal; Infant, Newborn; Genetic Diseases, Inborn
MeSH Terms: conditions — Disease; Genetic Diseases, Inborn

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention): Patients in this arm receive standard genetic evaluation without the addition of next generation sequencing for the diagnosis of their presumed genetic condition
- Rapid whole genome sequencing (StatSeq) (Experimental): Patients in this arm will receive standard of care genetic evaluation and next generation sequencing of their genome to achieve rapid diagnosis of genetic conditions.
  Interventions: Other: Rapid whole genome sequencing (StatSeq)

INTERVENTIONS:
Other: Rapid whole genome sequencing (StatSeq) — Patients in this arm will received standard genetic testing, the Perkins Elmer StepOne expanded newborn screen and the rapid whole genome sequencing (StatSeq). the receipt of the StatSeq testing is the different factor between arms. the standard genetic testing includes any testing that is clinically available to the attending physician that would normally be ordered for the patient if not enrolled in this study.
  Arms: Rapid whole genome sequencing (StatSeq)

SUMMARY:
The purpose of this study is to compare the effectiveness of rapid next generation sequencing (NGS, such as whole genome sequencing1) with current practice to provide diagnostic or prognostic information or treatment guidance in acutely ill neonates and infants, particularly with respect to clinical care, cost and outcomes.

DETAILED DESCRIPTION:
This is a randomized, blinded, prospective study examining the comparative effectiveness - both clinical and cost effectiveness - of rapid NGS (StatSeq), compared to standard of care, including an expanded newborn screen, in acutely ill neonates and infants with potential genetic diseases. Acutely ill neonates and infants who have an undiagnosed illness, and their families, will be eligible to participate in the study. The investigators will enroll approximately 1,000 neonates and infants at a single study site. The study population will be recruited from Children's Mercy Hospital inpatient population, primarily the intensive care nursery (ICN, also known as the NICU), with a smaller subpopulation presenting to other hospital services, such as the pediatric intensive care unit (PICU). All affected study participants will receive an expanded newborn screen (NBS). Newborn screening is biochemical testing of a heel-prick blood spot that is federally mandated to be performed on all US live births. 67 diseases are tested for by NBS in MO, most of which are genetic diseases. The expanded NBS proposed herein is the clinically available StepOne Newborn Screen® from Perkin Elmer, and will be performed in addition to standard State of MO screening on all enrolled infants in both arms. Half of the affected study participants will be randomized to receive StatSeq in addition to standard testing for their acute illness and expanded NBS. Additionally, all willing clinical providers will be enrolled and their perceptions on clinical outcomes will be measured.

All subjects will have blood drawn for nucleic acid (DNA and RNA) isolation and the expanded NBS at the time of enrollment in the study. All blood sample volumes will adhere to the CMH policy on maximum blood in pediatric patients. If the volume allowed for in this policy exceeds 5ml, 5 ml will be the maximum collected at enrollment. Buccal smears, heel-prick blood spots, additional blood, urine and tissue samples may be collected, if available as sample retains from other studies, and stored in the Center for Pediatric Genomic Medicine (CPGM) per their approved IRB protocol (IRB Study #11120514). The latter samples will not involve invasive sampling. Nucleic acids will be isolated and prepared for NGS with standard protocols at the CPGM (Center for Pediatric Genomic Medicine). Familial samples (for example, mother, father, affected or unaffected siblings) will also be obtained, and nucleic acids will also be sequenced per the Genome Center Biorepository protocol, as indicated, to assist in diagnosis of the acute medical condition in the newborn. All sequencing data will be stored in the Genome Center Biorepository (IRB Study #11120514).

A minimum of two expert Center data analysts will be responsible for analyzing the DNA variants following NGS. One of the analysts will then compile a report to be presented to the Molecular Pathology Laboratory Director or Assistant Director. In the case of positive study findings that may be diagnostic, the Molecular Pathology Laboratory Director or Assistant Director will perform confirmatory clinical diagnostic testing and, if confirmed, a standard clinical diagnostic report will be placed in the patient's medical record. In the case of acutely material (actionable) positive study findings, the results will be verbally conveyed to the primary clinical team directly prior to confirmatory testing. A generic research note will be placed in the patient's medical record that indicates that a verbal, provisional report was issued (Appendix A). Verbal, provisional reporting of results before confirmatory testing will only be performed in cases where the delay in reporting necessary for confirmation was likely to result in significant harm to the patient. Confirmatory testing will be performed promptly in all cases, including those in which in which a verbal report has been given. A case conference format may be utilized for return of results if the complexity of the diagnosis or potential treatment for that diagnosis warrants detailed discussion. If no potentially pathogenic variants are identified, a verbal report will be provided to the clinical care physician of record to communicate that there were no causative findings, and a generic research note will be placed in the medical record that states that nondiagnostic research grade NGS was performed (Appendix B). No negative diagnostic written report of results will be placed in the patient's chart in this instance, as there is no available clinical grade testing to confirm negative results for all genes tested. Follow up with the patient's family will be guided by the clinical care team. All study participants and their clinicians will be notified of randomization assignment at/by day 10 after randomization. This information will help alleviate anxiety on the part of the family, and also provides a mechanism for patient crossover into the rapid NGS arm if the patient is clinically deteriorating, and at the clinical care team's request. Rarely, those participants and clinicians will be notified sooner if they were randomized to the rapid NGS group and a diagnosis is made in less than 10 days. Both molecular diagnoses made and time to diagnosis will be recorded as primary outcomes.

All positive results from the Perkin Elmer StepOne expanded NBS (received by all enrolled infants and NOT a study variable) will be returned to the Genome Center personnel. Based on these results, confirmatory testing through Perkin Elmer will be performed if this condition was not identified on the standard State NBS screen for each infant. These provisional results will be verbally communicated with the primary clinician team and additional samples requested, if necessary, for confirmation. Upon confirmation, the results will be entered in the patient's medical record.

Each time a study participant is enrolled, the primary clinical providers will be asked to fill out a survey prior to StatSeq testing and after return of results. We will also review the patient's medical record and collect clinical variables including laboratory testing, radiology results, medications and other treatments received to further analyze the effect rapid NGS has on clinical care. We plan to follow up with families annually up to 5 years post enrollment and record clinical outcomes related to this study.

This study will be integrated with two other study protocols, one being the CMH Genomic Medicine Repository (IRB 11120514) and the other Genomes in newborns (#13120442) that studies the ethical and legal implications of rapid NGS in this population. Data records will be requested from both studies. The participants must agree to enroll in the Genome Center Biorepository. The Genomes in newborns study will be optional.

ELIGIBILITY:
Inclusion Criteria: One of the following criteria required.

* Clinical genetic testing or a genetic consult is ordered
* Subject has one major structural anomaly or three or more minor anomalies
* Abnormal laboratory testing suggestive of a genetic disease
* Abnormal response to standard therapy for a major underlying condition

Exclusion Criteria:

* Previously confirmed genetic diagnosis that explains the clinical condition
* Has features pathognomonic for a large chromosomal aberration (Trisomy 13, 18, 21 or other)

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Molecular Diagnosis Made | 28 days
  If randomized to the Rapid Genome Sequencing group, did the testing result in a molecular diagnosis for the patient with three weeks of receipt of the DNA in the lab.
Time to Molecular Diagnosis | 28 days
  How many days from enrollment were required in our to achieve a molecular diagnosis in the infant
Change in Clinical Management | 28 days
  If randomized to the Rapid Genome Sequencing group and a molecular diagnosis achieved, did it provide a change in clinical management as determined by a survey of primary care team attending via a survey

SECONDARY OUTCOMES:
Number of Consults | 28 days
  Total number of consultations including follow up required during hospitalization
Cost Effectiveness | 28 days
  Determination of utilization of healthcare resources in hospital charges in both arms

OTHER OUTCOMES:
Length of Stay | After 12 months
  Length of stay in days to discharge.
Number of Deaths | After 12 months
  Number of deaths in each group

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kingsmore, MB BAO ChB, Principal Investigator — Rady Children's Hospital; Steve Leeder, PhD, Principal Investigator — Children's Mercy Hospital and Clinics; Laurel K Willig, MD, Study Director — Children's Mercy Hospital and Clinics; Joshua E Petrikin, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States